CLINICAL TRIAL: NCT02751138
Title: Determination of Immune Phenotype in Glioblastoma Patients
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Andrej Pala, MD, University of Ulm
Other Study IDs: University Hospital Ulm
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Glioblastoma Multiforme
Keywords: Immune phenotype; Cytokines; Genetic aberration; Overall survival; Progression free survival
MeSH Terms: conditions — Glioblastoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cell (PBMC), Plasma, Tumor tissue, DNA, RNA, miRNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Isocitrate dehydrogenase - 1 mutated: Immunophenotype of Glioblastoma and correlation with outcome
  Interventions: Procedure: Surgery
- Isocitrate dehydrogenase - 1 wild type: Immunophenotype of Glioblastoma and correlation with outcome
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Tumor resection

SUMMARY:
Glioblastoma multiforme (GBM) is the most common primary brain tumor in adults. Despite intensive research efforts and a multimodal management that actually consists of surgery, radiotherapy and chemotherapy with temozolomide, the prognosis is dismal. The aim of the current observational study is to determine immune phenotypes in individual patients with GBM at the time of diagnosis and to correlate tumor size, location (imaging), tumor properties (isocitrate dehydrogenase - 1 (IDH-1), o6-methylguanine-DNA-methyltransferase (MGMT), epidermal growth factor receptor (EGFR) mutation status, etc.) with clinical data, such as progression free and overall survival, Karnofsky index (progression free survival (PFS),overall survival (OS), Karnofsky score( KFS)), with blood immune phenotypes, biomarkers, and immune histochemical results of tumor infiltrating lymphocytes, macrophages, myeloid derived suppressor cells (MDSC), etc.. The different immunological phenotypes could predict a positive response to specific immunological therapeutic strategies and select the individual therapeutic plan for an individual GBM patient.

ELIGIBILITY:
Inclusion Criteria:

* adult glioblastoma multiforme

Exclusion Criteria:

* pregnancy, unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult glioblastoma multiforme
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 months

SECONDARY OUTCOMES:
Progression free survival | 3 months
Karnofsky performance score | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Yes
Immune phenotypes of glioma patients included and clinical follow-up